CLINICAL TRIAL: NCT07069894
Title: Effect of Xuebijing InjecTion on Outcomes in Sepsis Patients Under Real-World Conditions: A Patient Registry
Brief Title: Effect of Xuebijing InjecTion on Outcomes in Sepsis Patients Under Real-World Conditions（EXIT-SEP REAL）
Acronym: EXIT-SEP REAL
Status: Not yet recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Songqiao Liu, Prof, Southeast University, China
Other Study IDs: 2025ZDSYLL252-P01
Record Dates: First submitted 2025-06-30; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Sepsis
Keywords: Sepsis; Xuebijing injection; Intensive Care Unit
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Xuebijing Group: The Xuebijing group consisted of sepsis patients who received both Xuebijing injection and guideline-concordant therapy. Researchers did not provide any additional interventions, but instead observed and documented the clinical outcomes and treatment effects of Xuebijing injection in combination with standard therapy.

SUMMARY:
Xuebijing injection (XBJ) showed proven efficacy in the EXIT-SEP trial (NCT03238742), lowering 28-day mortality. However, its real-world effectiveness requires validation due to the trial's strict criteria. Broader clinical evaluation is imperative.

DETAILED DESCRIPTION:
Sepsis is a life-threatening syndrome caused by a dysregulated response to infection, affecting an estimated 49 million people and claiming 11 million lives globally each year. Xuebijing injection (XBJ) has demonstrated efficacy in improving outcomes. A large multicenter randomized controlled trial (EXIT-SEP) confirmed that XBJ significantly reduces 28-day mortality. However, the trial population was relatively selected (aged 18-75 years, SOFA score 2-13), leaving its effectiveness in complex, real-world settings unclear. Therefore, further investigation of XBJ's impact in broader clinical practice is essential.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged ≥18 years
* Sepsis diagnosis meeting Sepsis-3 criteria
* Informed consent signed by patient or legally authorized representative

Exclusion Criteria:

* Patients with a prior history of sepsis
* Sepsis diagnosis >48 hours prior to enrollment
* Current participation in clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with sepsis (Sepsis-3 criteria) upon ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | 28 days after enrollment

SECONDARY OUTCOMES:
ICU mortality | From Intensive Care Unit (ICU) admission to ICU discharge or death, up to 28 days.
Ventilator-free days | 28 days after enrollment
ICU-free days within 28 days | 28 days after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ma Q, Qiu M, Zhou H, Chen J, Yang X, Deng Z, Chen L, Zhou J, Liao Y, Chen Q, Zheng Q, Cai L, Shen L, Yang Z. The study on the treatment of Xuebijing injection (XBJ) in adults with severe or critical Corona Virus Disease 2019 and the inhibitory effect of XBJ against SARS-CoV-2. Pharmacol Res. 2020 Oct;160:105073. doi: 10.1016/j.phrs.2020.105073. Epub 2020 Jul 9. No abstract available. PMID 32653650
- [Background] Liu X, Song Y, Guan W, Qiu H, Du B, Li Y, Liu Y, Shang H, Zhong N, Coronavirus Disease Emergency Project Research Collaboration G. [A multicenter prospective cohort study of Xuebijing injection in the treatment of severe coronavirus disease 2019]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2021 Jul;33(7):774-778. doi: 10.3760/cma.j.cn121430-20210514-00714. Chinese. PMID 34412743
- [Background] Song Y, Yao C, Yao Y, Han H, Zhao X, Yu K, Liu L, Xu Y, Liu Z, Zhou Q, Wang Y, Ma Z, Zheng Y, Wu D, Tang Z, Zhang M, Pan S, Chai Y, Song Y, Zhang J, Pan L, Liu Y, Yu H, Yu X, Zhang H, Wang X, Du Z, Wan X, Tang Y, Tian Y, Zhu Y, Wang H, Yan X, Liu Z, Zhang B, Zhong N, Shang H, Bai C. XueBiJing Injection Versus Placebo for Critically Ill Patients With Severe Community-Acquired Pneumonia: A Randomized Controlled Trial. Crit Care Med. 2019 Sep;47(9):e735-e743. doi: 10.1097/CCM.0000000000003842. PMID 31162191
- [Background] Liu S, Yao C, Xie J, Liu H, Wang H, Lin Z, Qin B, Wang D, Lu W, Ma X, Liu Y, Liu L, Zhang C, Xu L, Zheng R, Zhou F, Liu Z, Zhang G, Zhou L, Liu J, Fei A, Zhang G, Zhu Y, Qian K, Wang R, Liang Y, Duan M, Wu D, Sun R, Wang Y, Zhang X, Cao Q, Yang M, Jin M, Song Y, Huang L, Zhou F, Chen D, Liang Q, Qian C, Tang Z, Zhang Z, Feng Q, Peng Z, Sun R, Song Z, Sun Y, Chai Y, Zhou L, Cheng C, Li L, Yan X, Zhang J, Huang Y, Guo F, Li C, Yang Y, Shang H, Qiu H; EXIT-SEP Investigators. Effect of an Herbal-Based Injection on 28-Day Mortality in Patients With Sepsis: The EXIT-SEP Randomized Clinical Trial. JAMA Intern Med. 2023 Jul 1;183(7):647-655. doi: 10.1001/jamainternmed.2023.0780. PMID 37126332
- [Background] Xie J, Wang H, Kang Y, Zhou L, Liu Z, Qin B, Ma X, Cao X, Chen D, Lu W, Yao C, Yu K, Yao X, Shang H, Qiu H, Yang Y; CHinese Epidemiological Study of Sepsis (CHESS) Study Investigators. The Epidemiology of Sepsis in Chinese ICUs: A National Cross-Sectional Survey. Crit Care Med. 2020 Mar;48(3):e209-e218. doi: 10.1097/CCM.0000000000004155. PMID 31804299
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338